CLINICAL TRIAL: NCT05830344
Title: Evaluation of the Effect of Multi Radiance Medical® Super Pulsed Laser for Adjunctive Use in Providing Temporary Relief of Chronic Knee Pain of Musculoskeletal Origin
Brief Title: Effects of Multi Radiance Medical® Super Pulsed Laser on Chronic Knee Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Collaborators: Multi Radiance Medical (Industry)
Responsible Party: Principal Investigator, Ernesto Cesar Pinto Leal Junior, Full professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5.767.644
Record Dates: First submitted 2023-03-31; First posted 2023-04-26 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Knee Pain Chronic
Keywords: Photobiomodulation Therapy; LLLT

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A researcher will program the device (placebo or active) and will be instructed not to inform the patients or other researchers as to the type of treatment (placebo or active). Therefore, the researcher responsible for the treatment, the investigator and the outcome assessor will be blinded to the type of treatment being administered to the patients. The sounds and signals emitted from the device as well as the information displayed on the screen will be identical, regardless of the type of treatment (placebo or active).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo treatment will be irradiated using a Multi Radiance Medical Super Pulsed Laser, manufactured by Multi Radiance Medical® (Solon,Ohio, USA), at 5 sites in the knee area, without any emission of therapeutic dose. The treatment will be performed 3 times a week, for four consecutive weeks, yielding 12 treatments. The sounds and signals emitted from the device as well as the information displayed on the screen will be identical, regardless of the type of treatment (active or placebo).
  Interventions: Device: Placebo Multi Radiance Medical® Super Pulsed Laser
- Active (Experimental): Active treatment will be irradiated using a Multi Radiance Medical Super Pulsed Laser, manufactured by Multi Radiance Medical® (Solon,Ohio, USA), at 5 sites in the knee area, with a dose of 8.02 J per site. The treatment will be performed 3 times a week, for four consecutive weeks, yielding 12 treatments.
  Interventions: Device: Active Multi Radiance Medical® Super Pulsed Laser

INTERVENTIONS:
Device: Placebo Multi Radiance Medical® Super Pulsed Laser — Placebo, without therapeutic dose.
  Arms: Placebo
Device: Active Multi Radiance Medical® Super Pulsed Laser — Active with a dose of 8.02 J per site.
  Arms: Active

SUMMARY:
Knee pain is among the most common reasons for musculoskeletal pain consultations, accounting for nearly 4 million primary care visits annually. Knee pain can have different causes such as, tendinopathies, synovitis, bursitis, trauma, etc.

Considering the importance and high incidence of musculoskeletal disorders that affect the knee joint, a variety of therapeutic modalities has been employed to alleviate pain and repair the tissue. Among these conservative treatments, photobiomodulation therapy (PBMT) has been shown to stimulate tendon and ligament healing, and decrease the pain.

Therefore, the aim of this study is to determine the effectiveness of the Multi Radiance Medical® Super Pulsed Laser, manufactured by Multi Radiance Medical®, for adjunctive use in providing temporary relief of chronic knee pain of musculoskeletal origin.

DETAILED DESCRIPTION:
To achieve the proposed objectives it will be performed a randomized, triple-blind (patients, therapists, outcome assessors), placebo-controlled trial, with voluntary patients with chronic knee pain. Eighty-six patients will be randomly allocated to two treatment groups: 1. Active Multi Radiance Medical® Super Pulsed Laser or Placebo Multi Radiance Medical® Super Pulsed Laser. The patients will be treated by a blinded therapist.

Treatment administration will be performed 3 times a week, for four consecutive weeks, yielding 12 treatments (each treatment administration one to two days apart).

The outcomes will be obtained at the stabilization phase, baseline (pre-procedure), end of treatment and one week after the conclusion of treatment.

The data will be collected by a blinded assessor. The statistical analysis will follow the intention-to-treat principles.

The project was also approved by the Research Ethics Committee from Universidade Nove de Julho, under the number 5.332.202. Board Affiliation: Comissão Nacional de Ética em Pesquisa (CONEP) Phone: +55113385-9010 - Email: comitedeetica@uninove.br Address: Vergueiro nº 235/249. Liberdade, Sao Paulo, Sao Paulo, Brazil.

The investigators will analyze: degree of pain, levels of prostaglandin E2, subjective knee evaluation, patient satisfaction, blinded efficacy and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent form.
* Aged between 18 and 50 years, inclusive.
* Any gender.
* Subject is fluent in Portuguese.
* The volunteers' presenting primary (dominant) pain is in the region of the right or left knee only. i.e., it is unilateral.
* Self-reported degree of pain rating on the 0-100 VAS pain scale for the target knee is 50 or greater.
* Self-reported degree of pain rating on the 0-100 VAS pain scale for the non-target knee is less than 20.
* Knee pain is episodic chronic, defined as having occurred and recurred over regular or irregular periods or intervals of time, persisting over at least the last 3 months.
* Volunteers' knee pain is of benign musculoskeletal origin wherein the etiology is tendinopathies, synovitis, bursitis, strain, and sprain, of traumatic or non-traumatic origin, as determined by the principal investigator based on any one or combination of the following:
* Prior diagnosis by a qualified licensed medical professional current within the last 2 years evidenced through source documentation.
* Previous Records Review, such as x-ray, MRI, CT scans, etc., where available, that indicate muscle or ligament injury and the absence of Degenerative Joint Disorder (DJD).
* Medical history consistent with one of the etiologies of knee pain falling within the scope of this study.
* Physical examination of the knee that yields one or both of the following findings: Increased pain upon range of motion and/or increased pain and weakness upon knee extension, knee flexion, or gait.
* Subject is willing and able to maintain his or her individualized pain regimen as determined by the study principal investigator at baseline as needed to manage any knee pain that may arise throughout the course of study duration, whilst refraining from consuming other over the counter and/or prescription medication(s) and/or herbal supplements intended for the relief of pain and/or inflammation, and/or partaking in other treatments/therapies.

Exclusion Criteria:

A volunteer who satisfies any one or more of the following criteria will be excluded from study participation:

* The volunteers' presenting primary pain is located outside or in addition to the knee.
* The volunteers' presenting primary pain is bilateral, i.e., equally dominant in the right and left knees.
* Self-reported degree of pain rating on the 0-100 VAS pain scale for the target knee is less than 50.
* Self-reported degree of pain rating on the 0-100 VAS pain scale for the non-target knee is 20 or greater.
* Knee pain is acute, defined as having persisted less than half the time over less than the last 3 months.
* Knee pain is not episodic, such that it has either been continually present without respite over the past 3 months and/or there has not been recurrent episodes within the past 3 months.
* Volunteers' knee pain is of other than, or in addition to, benign musculoskeletal origin wherein the etiology is tendinopathies, synovitis, bursitis, strains, and sprains from traumatic or non-traumatic origin, and/or the etiology of the subject's knee pain cannot be satisfactorily ruled out.
* Prior surgical intervention to the target knee that in the opinion of the principal investigator may affect the study treatment and or outcomes assessment.
* Neurologic deficits that in the opinion of the principal investigator may affect the study treatment and or outcomes assessment.
* Peripheral nerve disease.
* Rheumatoid arthritis.
* Hip or ankle disease.
* Congenital or acquired bony deformity in the ipsilateral lower extremity.
* Secondary orthopedic problems that in the opinion of the principal investigator may affect the study treatment and or outcomes assessment.
* Local corticosteroids and/or botulinum toxin (Botox®) injection for knee pain relief within 30 days prior to study enrollment.
* Treatments such as chiropractic care, and acupuncture within 30 days prior to study enrollment.
* Current, active chronic pain disease, such as chronic fatigue syndrome, fibromyalgia, endometriosis, inflammatory bowel disease, interstitial cystitis diabetic neuropathic pain,
* Current cancer or treatment for cancer in the past 6 months.
* Significant heart conditions including chronic heart failure (CHF) and implantable heart devices such as a pacemaker.
* Active infection, wound, or other external trauma to the areas to be treated with the PBMT.
* Medical, physical, or other contraindications for, or sensitivity to, light therapy.
* Pregnant, breast feeding, or planning pregnancy prior to the end of study participation.
* Female subject of childbearing age who is unwilling to engage in effective medical contraceptive use while sexually active during the study procedure administration phase.
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in past two years.
* Developmental disability or cognitive impairment that in the opinion of the principal investigator would preclude adequate comprehension of the informed consent form and/or ability to record the necessary study measurements.
* Any other medical condition or medication use that in the opinion of the principal investigator may affect the study treatment and or outcomes assessment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Degree of pain rating | 4 weeks (end of treatment).
  Degree of pain rating will be measured by 0-100 standardized Visual Analog Scale (VAS). Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Degree of pain rating | One-week after the conclusion of the treatment.
  Degree of pain rating will be measured by 0-100 standardized Visual Analog Scale (VAS). Higher scores mean worse outcome.
Levels of Prostaglandin E2 (PGE2) | 4 weeks (end of treatment) and one-week after the conclusion of the treatment.
  Levels of PGE2 will be measured by blood samples.
Subjective knee evaluation | 4 weeks (end of treatment) and one-week after the conclusion of the treatment.
  Subjective knee evaluation will be measured by the International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form consisting in 18 items and contains the following three domains: 1) symptoms, including pain, stiffness, swelling, locking/catching, and giving way; 2) sports and daily activities; and 3) current knee function and knee function prior to knee injury (not included in the total score). Scores range from 0 points (lowest level of function and highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Patient satisfaction | 4 weeks (end of treatment) and one-week after the conclusion of the treatment.
  Patient satisfaction will be measured by 1-item Likert Scale. The scale uses the following responses: very satisfied = 5; somewhat satisfied = 4; neither satisfied nor dissatisfied = 3; somewhat dissatisfied n=2; very dissatisfied =1. Highest scores indicates better satisfaction.
Blinding efficacy | 4 weeks (end of treatment) and one-week after the conclusion of the treatment.
  The blinding efficacy will be measured by the percentage of volunteers and outcome assessor who correctly perceived their procedure group assignment and the percentage of volunteers and outcome assessor who did not correctly perceive their procedure group .
Adverse events | 4 weeks (end of treatment) and one-week after the conclusion of the treatment.
  Adverse events will be measured by report.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Laboratory of Phototherapy and Innovative Technologies in Health, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be available on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available during five years after the study completion.
Access Criteria: All IPD that underlie results in a publication will be available on reasonable request.